CLINICAL TRIAL: NCT05120505
Title: Efficacy and Safety of Metformin in the Treatment of Fragile X Syndrome
Brief Title: Metformin in Children With Fragile X Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FXS2021_1.0
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Fragile X Syndrome; Metformin
MeSH Terms: conditions — Fragile X Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): The patients will be obtain Metformin starting from 50mg everyday to 1-2g per day for 6 months.
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): The patients will be obtain starch tablets starting from 50mg everyday to 1-2g per day for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — The patients in this group will be obtain Metformin starting from 50mg everyday at night, and gradually increase to maximum tolerable dose of 1-2g per day according to weights of patients for 6 months.
  Arms: Metformin group
Drug: Placebo — The patients in this group will be obtain starch tablets (which had same appearance and size comparing to Metformin) starting from 50mg everyday to 1-2g per day according to weights of patients for 6 months.
  Arms: Placebo group

SUMMARY:
This study is a controlled trial of metformin in children with fragile X syndrome(FXS). The age of FXS children range from 2 to 16 years old. Participants will be randomized in a double-blind design to either drug or placebo for 6-month period. The primary objectives are to assess metformin in treatment of behavior problems, cognitive and language with fragile X syndrome.

DETAILED DESCRIPTION:
This is a single-center study at the Children's Hospital of Fudan University for FXS patients aged 2 to 16 years inclusive. It is a randomized, double-blind, placebo-controlled trial of metformin.

Studies showed that there were pathogenically over activates of mTOR and MAPK/ERK pathways in FXS. Metformin, a guanidine derivative ,has been shown to reduce mTORC1 pathway activity in an AMPK-dependent manner and has also been shown to reduce MAPK pathway activity. Metformin treatments for FXS have been reported in animal experiments, some open label trials of metformin in FXS patients had been reported. Therefore, metformin has potential to rescue symptoms in children with FXS.

In this study, researchers hope to investigate the improvement effect of metformin on FXS symptoms such as behavior problems, cognition, language.

The intervention period is 6 months, follow-up visit at 1 year. The researchers will also assess the side effects of the study medication throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Genetic testing confirms the diagnosis of FXS
* Participate in the study with the informed consent of the guardian
* BMI>the 3rd percentile
* Not taking more than 2 therapeutic drugs
* Able to receive regular follow-up visits

Exclusion Criteria:

* Malnutrition
* Primary heart disease
* Severe infection or acute clinical illness
* Gastrointestinal, renal, or hepatic disease
* Previous history of lactic acidosis
* previous use of metformin intolerant
* Use of angiotensin converting enzyme inhibitors, use of anticoagulants, vitamin B12 deficiency, alcohol consumption
* Unstable systemic diseases other than FXS
* Changes in clinical medication

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of scores of Aberrant Behavior Checklist (ABC) | From baseline to the 6th month
  Difference on the scores of the ABC from baseline to the 6th month. ABC is a 58-item behavior scale ranked from 0("not a problem") to 3("severe problem") being the most severe for each item. 5 subscales include irritability, lethargy, stereotypy , hyperactivity and inappropriate speech. The same parent of patient will complete the checklist from baseline to 6th month. The global score changes of ABC will be measured as the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Y, Li D, Hu C, Tian Y, Lu P, Hagerman RJ, Xu X, Xu Q. Effects of Metformin on children with Fragile X Syndrome: a randomized, double-blind, placebo-controlled trial. Mol Autism. 2025 Nov 25;16(1):57. doi: 10.1186/s13229-025-00691-z. PMID 41291951